CLINICAL TRIAL: NCT06452381
Title: Towards Sustainable Food Systems: Allergenicity Assessment of Green Marine Macroalga Ulva sp.
Brief Title: Allergenicity Assessment of Green Marine Macroalga Ulva sp.
Status: Active, not recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Ronit Confino-Cohen, Prof, Ministry of Health, Israel
Other Study IDs: MMC-0207-21; 3-16052 (Other Grant/Funding Number: The Chief Scientist Fund, Ministry of Health)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the allergenic potential in humans, we will conduct a three-stage clinical trial.

In the first group, 20 healthy volunteers will be involved. All volunteers will be examined by an allergy specialist before enrolment to the study. After receiving informed consent, all volunteers will undergo an allergy skin test to the study seaweed proteins as well as to common allergens. Participants with a skin test showing sensitization will be excluded. Volunteers will be fed by 5 gram of the study seaweed 2 times a week, under supervision, for 6 weeks. After 6 weeks of feeding, skin tests will be repeated. All participants, will undergo an open oral food challenge after one month of avoidance of the study seaweed protein. Uneventful food challenge will rule out food allergy in a specific volunteer.

Second, the extension clinical phase will be conducted with 100 healthy volunteers. The inclusion, exclusion and study design will be similar to the pilot study.

The third phase will be conducted in a group of high-risk patients aimed to find the frequency of allergy to the study seaweed in high risk patients. Study population: 20 volunteers with high risk to seaweed food allergy. Inclusion criteria: Adults (>18 years old, males and females) with at least one of the following: Active atopic dermatitis or fish or sea food allergy. Study design will be similar to the pilot study.

DETAILED DESCRIPTION:
To determine the allergenic potential in humans, we will conduct a three-stage clinical trial. The length of each phase will be 3 months. Serum will be sampled from all the participants before and at the end of each phase.

In the first group, 20 volunteers will be involved. Inclusion criteria: Adults (>18); Males and females (10 males and 10 females) with no history of food allergy or atopy. Exclusion criteria: any history of food allergy, women pregnant or lactating, any history of atopy (moderate/severe atopic dermatitis, allergic rhinitis, asthma), any chronic diseases, any chronic medication use (except CP).

Study design: All volunteers will be examined by an allergy specialist before enrolment to the study to rule out any of the exclusion criteria. Volunteers with any of the exclusion criteria will be excluded from participation in this part of the study. After receiving informed consent, all volunteers will undergo an allergy skin test to the study seaweed proteins as well as to fish, sea foods , peanut, sesame, milk, soy, house dust mite and common Israeli pollens. Participants with a skin test showing sensitization by skin tests will be excluded from this part of the study. All volunteers passing the above stages will be enrolled. Volunteers will be fed by 5 gram of the study seaweed 2 times a week, under supervision, for 6 weeks. After 6 weeks of feeding, skin tests will be repeated. All participants, disregarding the results of the skin test, will undergo an open oral food challenge after one month of avoidance of the study seaweed protein. The open oral food challenge will include ingestion of 5 gram of the study seaweed protein and 2 hours of observation. An allergic reaction to the food challenge will be determined by the allergy specialist conducting the food challenge by predefined clinical signs and symptoms. If needed, first aid treatment will be provided by the allergy specialist. Uneventful food challenge will rule out food allergy in a specific volunteer. Expected results: we assume that the study seaweed is not more allergenic than other common foods. Thus, we expect that no more than one volunteer will have a reaction to the food challenge.

Second, the extension clinical phase will be conducted with 100 healthy volunteers. The sample size was based on the prevalence of IgE mediated food allergy (of all kinds) in the general population and engineering constraints for extraction process scale up. Finding at least one person with the allergy should be around 63% confidence under the prevalence of 1%, and 95% confidence under a prevalence of 3% and a sample size of 100. The inclusion, exclusion and study design will be similar to the pilot study. Blood test will be drawn from patients that will be found to be allergic to the seaweed in order to try to define specific allergenic epitopes of the seaweed. Expected outcomes: allergy to the study seaweed will be found in less than 5% of healthy volunteers.

The third phase will be conducted in a group of high-risk patients aimed to find the frequency of allergy to the study seaweed in high risk patients. Study population: 20 volunteers with high risk to seaweed food allergy. Inclusion criteria: Adults (>18 years old, males and females) with at least one of the following: Active atopic dermatitis or fish or sea food allergy. Study design will be similar to the pilot study. Blood tests will be drawn from patients that will be found to be allergic to the seaweed in order to try and define specific allergenic epitopes of the seaweed. We expect that allergy to the study seaweed protein will be found in less than 10% of high-risk volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18)
* Males and females (10 males and 10 females) with no history of food allergy or atopy

Exclusion Criteria:

* Any history of food allergy, women pregnant or lactating, any history of atopy (moderate/severe atopic dermatitis, allergic rhinitis, asthma), any chronic diseases, any chronic medication use (except CP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
An allergic reaction to the food challenge | 10 weeks
  After 6 weeks of repeated eating All participants, disregarding the results of the skin test, will undergo an open oral food challenge after one month of avoidance of the study seaweed protein. The open oral food challenge will include ingestion of 5 gram of the study seaweed protein and 2 hours of observation. An allergic reaction to the food challenge or its absence is the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Derived] Kedar O, Golberg A, Obolski U, Steinbruch E, Chemodanov A, Israel A, Livney YD, Lachover-Roth I, Rosman Y, Confino-Cohen R. Initial allergenicity assessment of Ulva sp. seaweed flour. NPJ Sci Food. 2025 Dec 3;10(1):1. doi: 10.1038/s41538-025-00638-x. PMID 41339625